CLINICAL TRIAL: NCT04200092
Title: A Two Part Study Investigating the Safety and pk of Single Ascending Doses of Staccato Granisetron (AZ-010) and Crossover Comparison of the Pharmacokinetics and Safety of AZ-010 and Intravenous Granisetron in Healthy Volunteers
Brief Title: Staccato® Granisetron Single Dose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMDC-010-101
Record Dates: First submitted 2019-11-20; First posted 2019-12-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Granisetron; Equipment and Supplies; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Part A: Cohort 1 (Experimental): A single oral dose of 0.5 mg AZ-010 (Staccato Granisetron) administered to 8 subjects, with at least 2 males and 2 females. Each subject received a single dose of 0.5 mg AZ-010, or matching Staccato® placebo; 6 subjects received AZ-010 and 2 subjects received Staccato® placebo.
  Upon completion of the cohort, a review of the in-clinic safety and tolerability data was performed by the PI, Medical Monitor, and an independent data safety monitoring board (DSMB) to determine if there were adequate safety and tolerability data to support escalation to the next dose. Safety was evaluated by the PI, Medical Monitor, and DSMB upon completion of Part A and prior to start of Part B.
  Each subject participated for up to 4 weeks, depending upon the timing of screening.
  Subjects were confined to the clinic for 4 days (3 nights). A follow-up phone call was conducted, approximately 7 days after the subject left the CRU.
  Interventions: Combination Product: 0.5mg AZ-010; placebo
- Part A: Cohort 2 (Experimental): A single oral dose of 1 mg AZ-010 (Staccato Granisetron) administered to 8 subjects, with at least 2 males and 2 females. Each subject received a single dose of 1 mg AZ-010, or matching Staccato® placebo; 6 subjects received AZ-010 and 2 subjects received Staccato® placebo.
  Upon completion of the cohort, a review of the in-clinic safety and tolerability data was performed by the PI, Medical Monitor, and an independent data safety monitoring board (DSMB) to determine if there were adequate safety and tolerability data to support escalation to the next dose. The single daily dose did not exceed 3 mg. Safety was evaluated by the PI, Medical Monitor, and DSMB upon completion of Part A and prior to start of Part B.
  Each subject participated for up to 4 weeks, depending upon the timing of screening.
  Subjects were confined to the clinic for 4 days (3 nights). A follow-up phone call was conducted, approximately 7 days after the subject left the CRU.
  Interventions: Combination Product: 1mg AZ-010
- Part A: Cohort 3 (Experimental): A single oral dose of 3 mg AZ-010 (Staccato Granisetron) administered to 8 subjects, with at least 2 males and 2 females. Each subject received a single dose of 3 mg AZ-010, or matching Staccato® placebo; 6 subjects received AZ-010 and 2 subjects received Staccato® placebo.
  Upon completion of the cohort, a review of the in-clinic safety and tolerability data was performed by the PI, Medical Monitor, and an independent data safety monitoring board (DSMB) to determine if there were adequate safety and tolerability data to support escalation to the next dose. The single daily dose did not exceed 3 mg. Safety was evaluated by the PI, Medical Monitor, and DSMB upon completion of Part A and prior to start of Part B.
  Each subject participated for up to 4 weeks, depending upon the timing of screening.
  Subjects were confined to the clinic for 4 days (3 nights). A follow-up phone call was conducted, approximately 7 days after the subject left the CRU.
  Interventions: Combination Product: 3mg AZ-010
- Part B: Sequence 1 (Active Comparator): A single inhalation dose of 1 mg AZ-010, followed by IV injection granisetron 1mg, 2-period, a 2-treatment open-label crossover design.
  Participants were randomized in a 1:1 ratio to 1 of 2 sequences. Period 1 began with the inhalation dose of AZ-010 1mg and after a three-day washout participants were crossed over to the other sequence for Period 2 with the treatment of IV injection granisetron 1 mg dose.
  There was a total of 12 subjects (6 subjects in each sequence, with at least 2 males and 2 females in each sequence). Sequence 1 participants crossed over to Sequence 2 after washout.
  Interventions: Combination Product: AZ-010 1mg; Drug: IV Granisetron 1mg
- Part B: Sequence 2 (Active Comparator): Treatment of 1 mg (IV) granisetron followed by a single inhalation dose of AZ-010 1mg, a 2-period, 2-treatment open-label crossover design.
  Part B Sequence 2 participants began with Period 1 treatment of IV injection granisetron 1 mg dose and after a three-day washout participants were crossed over to the other sequence for Period 2 with the inhalation dose of AZ-010 1mg.
  There was a total of12 subjects (6 subjects in each sequence, with at least 2 males and 2 females in each sequence). Sequence 2 participants crossed over to Sequence 1 after washout.
  Interventions: Combination Product: AZ-010 1mg; Drug: IV Granisetron 1mg
- Pooled Placebo, Cohort 1, 2, 3 Part A (Placebo Comparator): Participants in Part A, Cohorts 1, 2, and 3, double-blind, randomized, and placebo-controlled study who received placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: 0.5mg AZ-010; placebo — Subject will receive a single inhaled dose (0.5mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Granisetron 0.5 mg
  Arms: Part A: Cohort 1
Combination Product: 1mg AZ-010 — Subject will receive a single inhaled dose (1.0 mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Granisetron 1mg
  Arms: Part A: Cohort 2
Combination Product: 3mg AZ-010 — Subject will receive a single inhaled dose (3.0 mg) of AZ-010 or matching Staccato Placebo
  Other Names: Staccato Granisetron 3mg
  Arms: Part A: Cohort 3
Combination Product: AZ-010 1mg — 2-period, 2-treatment open-label crossover design
  Other Names: Staccato Granisetron 1mg
  Arms: Part B: Sequence 1; Part B: Sequence 2
Drug: IV Granisetron 1mg — 2-period, 2-treatment open-label crossover design
  Other Names: Granisetron HCl, supplied as a 1 mg/mL solution (Lot No. 061488A)
  Arms: Part B: Sequence 1; Part B: Sequence 2
Other: Placebo — Participants in Part A, Cohorts 1, 2, and 3, double-blind, randomized, and placebo-controlled study who received placebo.
  Arms: Pooled Placebo, Cohort 1, 2, 3 Part A

SUMMARY:
This study was conducted in 2 parts in separate treatment groups of healthy volunteers. Part A of the study was double-blind, randomized, and placebo-controlled; Part B is open label.

The primary objectives for each part were as follows:

Part A:

1. To examine the tolerability and safety of single ascending doses up to 3 mg of AZ-010 (Staccato Granisetron) in healthy volunteers
2. To characterize the pharmacokinetics (PK) of single ascending doses up to 3 mg of AZ-010 in healthy volunteers

Part B:

1. To compare the PK and safety of a single dose of 1 mg of AZ-010 with that of 1 mg granisetron hydrochloride intravenous (IV) injection in healthy volunteers.

The 2 parts to the study were performed sequentially.

DETAILED DESCRIPTION:
Part A assessed single ascending orally inhaled doses of AZ-010 in a double-blind, placebo controlled design. The planned AZ-010 doses to be studied were 0.5 mg, 1 mg, and 3 mg delivered from 1 device each.

There were 3 cohorts of at least 8 subjects each, with at least 2 males and 2 females in each cohort. Each subject received a single dose of AZ-010, or matching Staccato® placebo; 6 subjects received AZ-010 and 2 subjects received Staccato® placebo per cohort.

Upon completion of each cohort, a review of the in-clinic safety and tolerability data was performed by the Principal Investigator (PI), Medical Monitor, and an independent data safety monitoring board (DSMB) to determine if there were adequate safety and tolerability data to support escalation to the next dose up to 3 mg.

Safety was evaluated by the PI, Medical Monitor, and DSMB upon completion of Part A and prior to start of Part B. PK data were analyzed and assessed through blood samples obtained for Parts A and B.

Part B Approximately 12 healthy volunteers were enrolled in this 2-period, 2-treatment open-label crossover design study assessing the PK profiles of AZ-010 (1 mg) and IV granisetron (1 mg).

Eligible consenting subjects were randomized to 1 of 2 treatment sequences, with a total of 12 subjects (6 subjects in each sequence, with at least 2 males and 2 females in each sequence).

Treatment periods were separated by at least a 3-day washout between doses.

ELIGIBILITY:
Inclusion Criteria

1. Healthy adult males and females between 18 and 60 years of age, inclusive at the time of signing the informed consent document.
2. Female subjects fulfilled the following criteria:

   1. Surgically sterile (including bilateral tubal ligation) for at least 3 months prior to screening
   2. Postmenopausal, defined as 1 of the following:

      * Last menstrual sequence greater than 12 months prior to screening
      * Last menstrual sequence greater than 6 months prior to screening and a serum follicle-stimulating hormone (FSH) concentration > 40 mIU/mL
   3. Subjects of childbearing potential (i.e., did not meet the criteria for surgical sterility or post- menopausal status outlined above):

      * Had a negative serum pregnancy test at screening and Day -1, as verified by the study doctor prior to starting study therapy
      * Either committed to true abstinence from heterosexual contact or agreed to use, and was able to comply with, effective contraception without interruption with one of the following methods during the study participation up until 90 days after administration of study drug: Oral contraceptive medications, Intrauterine devices, Hormonal implants, Injectable contraceptive medications, Double barrier methods.
3. Male subjects practiced true abstinence from heterosexual contact or, during sexual contact with a pregnant female or a female of childbearing potential, agreed to use a condom.
4. Healthy, as determined by the responsible physician, based on a medical evaluation including history, physical examination, vital signs, ECGs, and laboratory tests assessed at the screening visit and prior to the first dose of study drug.
5. Body weight ≥ 50 kg and BMI within the range of 18 to 32 kg/m2, inclusive, at screening.
6. Negative urine tests for selected drugs of abuse and alcohol breath test at screening and Day 1.
7. Dietary habits that fell within the range of normal, as determined by the PI.
8. Was willing and able to be confined at the clinical research center for the study period, and adhered to overall study visit schedule, procedures and other protocol requirements.
9. Understood and voluntarily signed an ICF prior to any study related assessments/procedures being conducted.

Exclusion Criteria

Subject candidates were not enrolled in the study if they met any of the following criteria:

1. Any significant medical condition, psychiatric illness or history of depression that could have, in the PI's opinion, compromised the subject's safety or interfered with the completion of this study.
2. Any condition, including the presence of laboratory abnormalities or abnormal pulmonary function test, which according to the PI, placed the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that according to the PI confounded the ability to interpret data from the study such as a virus, seasonal allergy, concurrent skin rash, etc. at screening or prior to drug treatment phase that may have been difficult to discern from further health status changes from an investigational product.
4. History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary (e.g., asthma, chronic obstructive pulmonary disease), metabolic, renal, hepatic, or gastrointestinal (GI) conditions including gastric bypass or other weight loss surgical procedure; or history of such conditions that, in the opinion of the PI, may have placed the subject at an unacceptable risk as a participant in this trial, may have interfered with the interpretation of safety and/or tolerability data obtained in the trial, or may have interfered with the absorption, distribution, metabolism, or excretion of the study drugs.
5. Used drugs known to prolong the corrected QT interval (QTc).
6. PR interval > 220 msec or QRS duration > 120 msec or Fridericia's corrected QT interval (QTcF) > 450 msec for men and > 470 msec for women obtained at the screening visit or prior to the first dose of study drug.
7. Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), serum creatinine, or total bilirubin > 1.5 upper limit of normal (ULN) at screening or prior to the first dose of study drug.
8. Positive blood screen for HIV antibody, hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at screening.
9. History of drug or alcohol abuse within 6 months of screening.
10. History of any tobacco product use within 3 months prior to the study.
11. Participation in a clinical trial and receipt of an investigational medication or a new chemical entity within 90 days, 5 half-lives, if known, or twice the duration of the biological effect of any medication (whichever is longer) prior to the first dose of current study drug.
12. Use of non-prescription medications, including herbal and dietary supplements within 5 days or 5 half-lives (whichever was longer) prior to the first dose of study drug.
13. Use of any 5-HT3 receptor antagonists or any other serotonergic drugs, including selective serotonergic reuptake inhibitors (SSRIs) or serotonin and norepinephrine reuptake inhibitors (SNRIs) within 5 days or 5 half-lives (whichever is longer) prior to screening.
14. Consumption of any caffeine and/or xanthine products (i.e., coffee, tea, chocolate and caffeine containing sodas, colas, etc.) within 24 hours prior to entry to the clinical unit on Day -1.
15. Donation of blood, plasma, or other blood products or blood collection in excess of 470 mL within 8 weeks prior to dosing.
16. Known history of sensitivity to any of the study drugs or components thereof, or to other 5-HT3 receptor antagonists, or a history of medication allergy or other allergy that, in the opinion of the PI, contraindicated study participation.
17. Major surgery within 4 weeks of screening that could have interfered with, or for which the treatment might have interfered with, the conduct of the study, or that would have posed an unacceptable risk to the subject in the opinion of the PI.
18. Uncontrolled current illness (i.e., active infection).
19. Had current or a history of cancer, with the exception of basal cell carcinoma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 3 days
  Number of Subjects with Adverse Events as a Measure of Safety and Tolerability
Measurement of Granisetron Exposure in Plasma | 3 days
  AUC (area under the curve)
Measurement of Granisetron Maximum Exposure in Plasma | 3 days
  Cmax
Measurement of Granisetron Time to Maximum Exposure in Plasma | 3 days
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Mathew, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States